CLINICAL TRIAL: NCT01628952
Title: Comparison of the Bilateral Transversus Abdominis Plane (TAP) Block Versus Curare in Muscle Relaxation of the Abdominal Wall During Laparoscopic Digestive Surgery: Prospective Randomized Study
Brief Title: Comparison of the Bilateral TAP Block Versus Curare in Muscle Relaxation of the Abdominal Wall During Laparoscopic Digestive Surgery: Prospective Randomized Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI2012_843_0007; 2012-000673-23 (EudraCT Number)
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: The Main of This Study is to Compare the Nerve Block of the Muscles of the Abdominal Wall Between the Bilateral TAP Block and Curare
MeSH Terms: interventions — Curare

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP (Experimental)
  Interventions: Drug: Transversus Abdominis Plane
- curare (Active Comparator): Patients will be randomized into two parallel groups. One group will receive curare, another benefit of a bilateral TAP block
  Interventions: Drug: Curare

INTERVENTIONS:
Drug: Transversus Abdominis Plane — PIA coelioscopic
  Arms: TAP
Drug: Curare — IAP coelioscopic
  Arms: curare

SUMMARY:
This is a Biomedical Research, prospective, randomized, controlled single-blind mono centric, phase IV comparison trial of the bilateral TAP block versus curare in muscle relaxation of the abdominal wall during laparoscopic digestive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and under 75 years
* Informed consent signed
* ASA I, II and III
* Patient affiliated to social security

Exclusion Criteria:

* ASA IV

  * BMI> 35 kg / m
  * Personal or family history of malignant hyperthermia
  * History of allergy or hypersensitivity to intravenous anesthetics (remifentanil), local anesthetics or muscle relaxants
  * Contraindications to sevoflurane: a history of malignant hyperthermia, history of liver disease after sevoflurane anesthesia, halogenated agents or hypersensitivity to any of these components.
  * Contraindications to succinylcholine: hyperkalemia, plasma cholinesterase deficiency nickname, para or tetraplegia more than 24 hours, burns over 24
  * Contraindications to cisatracurium: myasthenia
  * Neuromuscular diseases
  * Contraindications to local anesthetics: hypersensitivity to local anesthetics of the amide, intravenous regional anesthesia, porphyria, ventricular atrial conduction disturbances, epilepsy uncontrolled by treatment
  * Pregnancy and lactation
  * severe coagulation disorders
  * Inability to understand and give informed consent
  * Patient under guardianship, curatorship or protected
  * Indication of use of a hypnotic ketamine (BIS change)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Muscle relaxation. | 20 minutes after anesthesia induction
  Muscle relaxation of the abdominal wall will be evaluated based on the amount of volume infused initially to create the pneumoperitoneum. This parameter is given by the unit of laparoscopy and allow us to calculate the abdominal compliance (C = ΔV / Ap).

CONTACTS AND LOCATIONS:
Overall Officials: Hervé DUPONT, PU-PH, Study Director — CHU Amiens France
Locations (1):
- CHU Amiens, Amiens, Picardie, France

REFERENCES:
- [Result] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478